CLINICAL TRIAL: NCT01826422
Title: Effect of Eicosapentaenoic Fatty Acid (EPA) and Docosahexaenoic Fatty Acids (DHA) Supplementation on the Inflammation State and Metabolic Disorders in Patients With Duchenne Muscular Dystrophy or Becker Muscular Dystrophy
Brief Title: Effect of EPA and DHA in the Inflammation and Metabolic Disorders in DMD/DMB Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Nacional de Rehabilitacion (Other Government)
Responsible Party: Principal Investigator, Maricela Rodriguez Cruz, PhD, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DHA/EPA in Dunchenne; 180058 (Other Grant/Funding Number: CONACYT)
Record Dates: First submitted 2013-04-04; First posted 2013-04-08 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Muscular Dystrophy; Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Omega 3; Eicosapentaenoic fatty acid; Docosahexaenoic fatty acid
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPA and DHA (Experimental): Supplementation of 2.7 g/d of EPA and DHA were provided in 10 capsules per day (4 in the morning, 3 in the afternoon and 3 at night) during a period of 6 months. The capsules sizes were specially for children to improved the feeding process and its presentation is in gelatin capsules. The supplement is purified fish oil with pharmaceutical grade.
  Interventions: Dietary Supplement: EPA and DHA
- Placebo Comparator (Placebo Comparator): Supplementation of placebo with sunflower fatty at doses of 2.7 g/d were provided in 10 capsules per day (4 in the morning, 3 in the afternoon and 3 at night) during a period of 6 months. The capsules sizes are specially for children to improved the feeding process. This placebo is sunflower oil, so, it did not present anti-inflammatory or insulin sensitivity effects.
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: EPA and DHA — Each capsule contains 225mg of DHA, 45mg of EPA, other omega 3 fatty acids 20mg.
  Other Names: omega 3 fatty acid
  Arms: EPA and DHA
Dietary Supplement: Placebo Comparator — Placebo capsules will contain gelatin and sunflower oil. Fatty acid composition is as follows: lauric (C12:0), 0.19%; myristic (C14:0), 0.29%; palmitic (C16:0), 7.59%; palmitoleic (C16:1), 0.25%; stearic (C18:0), 3.49%; oleic (C18:1), 31.08%; linolenic (C18:3), 1.13%; linoleic (C18:2), 55.64%; DHA 0.02%; arachidic (C20:0), 0.30% and arachidonic (C20:4), 0.01%.
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to evaluate the effect of docosahexaenoic fatty acid and eicosapentaenoic fatty acid supplementation for six months on the inflammation state as well as the process of muscular regeneration and the metabolic disorders like obesity and insulin resistance in patients with Duchenne muscular dystrophy (DMD) and Becker muscular dystrophy (DMB) compared to those receiving placebo.

DETAILED DESCRIPTION:
DMD and DMB are X-linked diseases caused by mutations in the DMD gene, these mutations have important functional and structural consequences in skeletal muscle. In muscle fiber is observed inflammation and necrosis as a result of lost regenerative capacity. The muscle fibers can be replaced by connective and adipose tissue. In a previous study the investigators identified that 50% of Duchenne and Becker patients in the range of thirteen years old have obesity. In addition, these patients (N=66) have hyperinsulinemia (53.7%) and insulin resistance (48.5%). It is well known that obesity, hyperinsulinemia and insulin resistance have a inflammatory background.

It has been demonstrated that eicosapentaenoic fatty acid (EPA) and docosahexaenoic fatty acid (DHA) exhibit anti-inflammatory properties and have beneficial effects on obesity, hyperinsulinemia and insulin resistance in children and adolescents.

Objective: Determine the effect of EPA and DHA on inflammation, obesity and insulin resistance in patients with DMD/DMB compared to those receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and assent by the patient and both parents or guardian.
* Patients with clinical diagnosis of Duchenne Muscular Dystrophy (DMD) or Becker Muscular Dystrophy (DMB)
* Patients were not under treatment with corticosteroids

Exclusion Criteria:

* Patients decided to withdraw from the study
* Consumption of dietary supplements containing polyunsaturated fatty acids omega 3.
* With hypersensitivity to fish oil.
* Patients with respiratory and gastrointestinal problems. Medical responsible assessment the presence of respiratory and gastrointestinal problems.
* Patients with difficulty swallowing food, including those who have the difficulty ingesting oil capsules.
* Gastrostomy fed patients.

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maricela Rodriguez-Cruz, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Unit of Medical Researcha in Nutrition, Pediatric Hospital, IMSS., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz Guzman Odel R, Chavez Garcia AL, Rodriguez-Cruz M. Muscular dystrophies at different ages: metabolic and endocrine alterations. Int J Endocrinol. 2012;2012:485376. doi: 10.1155/2012/485376. Epub 2012 Jun 3. PMID 22701119
- [Background] Rodriguez-Cruz M, Sanchez R, Escobar RE, Cruz-Guzman Odel R, Lopez-Alarcon M, Bernabe Garcia M, Coral-Vazquez R, Matute G, Velazquez Wong AC. Evidence of Insulin Resistance and Other Metabolic Alterations in Boys with Duchenne or Becker Muscular Dystrophy. Int J Endocrinol. 2015;2015:867273. doi: 10.1155/2015/867273. Epub 2015 May 19. PMID 26089900
- [Result] Rodriguez-Cruz M, Cruz-Guzman ODR, Almeida-Becerril T, Solis-Serna AD, Atilano-Miguel S, Sanchez-Gonzalez JR, Barbosa-Cortes L, Ruiz-Cruz ED, Huicochea JC, Cardenas-Conejo A, Escobar-Cedillo RE, Yam-Ontiveros CA, Ricardez-Marcial EF. Potential therapeutic impact of omega-3 long chain-polyunsaturated fatty acids on inflammation markers in Duchenne muscular dystrophy: A double-blind, controlled randomized trial. Clin Nutr. 2018 Dec;37(6 Pt A):1840-1851. doi: 10.1016/j.clnu.2017.09.011. Epub 2017 Sep 23. PMID 28987470
- [Derived] Villaldama-Soriano MA, Rodriguez-Cruz M, Hernandez-De la Cruz SY, Almeida-Becerril T, Cardenas-Conejo A, Wong-Baeza C. Pro-inflammatory monocytes are increased in Duchenne muscular dystrophy and suppressed with omega-3 fatty acids: A double-blind, randomized, placebo-controlled pilot study. Eur J Neurol. 2022 Mar;29(3):855-864. doi: 10.1111/ene.15184. Epub 2021 Nov 26. PMID 34779542
- [Derived] Rodriguez-Cruz M, Atilano-Miguel S, Barbosa-Cortes L, Bernabe-Garcia M, Almeida-Becerril T, Cardenas-Conejo A, Del Rocio Cruz-Guzman O, Maldonado-Hernandez J. Evidence of muscle loss delay and improvement of hyperinsulinemia and insulin resistance in Duchenne muscular dystrophy supplemented with omega-3 fatty acids: A randomized study. Clin Nutr. 2019 Oct;38(5):2087-2097. doi: 10.1016/j.clnu.2018.10.017. Epub 2018 Oct 30. PMID 30420291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study were enrolled DMD/DMB patients from four Hospitals from Mexico city.
Groups:
- EPA and DHA: Patients received 2.9 g of EPA and DHA per day in 10 capsules (4 in the morning, 3 in the afternoon and 3 at night) during a period of 6 months. Each capsule contains 245mg of DHA, 45mg of EPA, other omega 3 50mg, oleic acid 60mg and Vitamin E 7.5 I. U
- Sunflower Oil: Patients received capsules of placebo sunflower fatty at doses of 10 capsules per day (4 in the morning, 3 in the afternoon and 3 at night) during a period of 6 months. The placebo capsules contain each gram contains: myristic (C14: 0 0) 1 mg, palmitic (C16: 0) 62mg, stearic (C18: 0) 43mg, palmitoleic (C16: 1) 1mg, oleic (C18: 1) 202mg, linolenic (C18: 3) 1mg and linoleic (C18: 2) 632mg
Period: Overall Study
Arm/Group | EPA and DHA | Sunflower Oil
Started | 18 | 22
Completed | 17 | 19
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EPA and DHA | Sunflower Oil | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 19 | 36
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.3 (3.1) | 8.6 (2.9) | 8.1 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 19 | 36
Region of Enrollment [Number; unit: participants]
  Mexico | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Body Composition (Body Fat)
Description: We observed changes in body composition such as total body fat by Dual X-ray Absorptiometry (DXA).
Time Frame: At baseline and at months 3 and 6 of supplementation.
Measure: Median (Full Range); unit: g/Kg of body weight
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
g/Kg of body weight
  Basal | 172.1 [84.7 to 530.4] | 232.7 [122.5 to 542.0]
  Month 3 after supplement | 180.2 [95.2 to 540.2] | 274.8 [124.4 to 547.3]
  Month 6 after supplement | 181.9 [98.0 to 535.0] | 298.2 [120.7 to 567.2]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

2. Primary Outcome: Lean Mass
Description: We observed changes in body composition such as total lean mass by Dual X-ray Absorptiometry (DXA).
Time Frame: At baseline and at months 1, 2, 3, 4, 5 and 6 of supplementation.
Measure: Mean (Full Range); unit: g/kg of body weight
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
g/kg of body weight
  Basal | 774.7 [429.1 to 857.3] | 662.4 [413.3 to 841.4]
  Month 1 after supplement | 769.6 [427.0 to 846.0] | 647.7 [420.4 to 827.6]
  Month 2 after supplement | 772.4 [419.9 to 851.5] | 630.6 [420.1 to 827.4]
  Month 3 after supplement | 757.7 [421.0 to 838.7] | 627.7 [414.5 to 835.2]
  Month 4 after supplement | 755.7 [416.9 to 855.0] | 605.7 [414.0 to 823.6]
  Month 5 after supplement | 768.6 [423.6 to 829.8] | 617.7 [433.0 to 811.6]
  Month 6 after supplement | 766.7 [426.2 to 849.9] | 606.2 [398.1 to 813.1]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

3. Primary Outcome: Anthropometric Measurement: Body Mass Index
Description: We measured weight, height by anthropometric to calculate the body mass index (body mass index).
Time Frame: At baseline and at months 1, 2, 3, 4, 5 and 6 of supplementation.
Measure: Median (Full Range); unit: g/m^2
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
g/m^2
  Basal | 42.5 [20.4 to 97.0] | 72.7 [1.8 to 98.4]
  Month 1 after supplement | 48.2 [9.6 to 97.2] | 78.3 [3.9 to 98.7]
  Month 2 after supplement | 49.6 [3.7 to 97.6] | 83.2 [5.4 to 98.5]
  Month 3 after supplement | 47.4 [15.3 to 97.2] | 82.2 [4.8 to 97.7]
  Month 4 after supplement | 49.9 [14.8 to 95.9] | 73.7 [9.8 to 98.0]
  Month 5 after supplement | 47.4 [3.4 to 96.5] | 75.3 [7.7 to 98.1]
  Month 6 after supplement | 51.7 [9.5 to 96.8] | 73.6 [5.3 to 98.2]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

4. Primary Outcome: Glucose in Serum
Description: A fasting blood sample was taken; serum glucose (mg/dL) levels were measured by the glucose-oxidase method.
Time Frame: At baseline and at months 1, 2, 3, 4, 5 and 6 of supplementation.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
mg/dL
  Basal | 83.5 [77.0 to 98.0] | 89.0 [76.0 to 121.0]
  Month 1 after supplement | 84.5 [79.0 to 98.0] | 90.0 [81.0 to 98.0]
  Month 2 after supplement | 87.5 [74.0 to 93.0] | 89.0 [79.0 to 107.0]
  Month 3 after supplement | 84.0 [61.0 to 95.0] | 86.8 [79.5 to 99.0]
  Month 4 after supplement | 83.0 [72.0 to 97.0] | 87.0 [82.0 to 107.0]
  Month 5 after supplement | 84.0 [76.0 to 99.0] | 89.8 [75.0 to 99.0]
  Month 6 after supplement | 82.0 [76.0 to 98.0] | 88.0 [78.0 to 99.0]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney) — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

5. Primary Outcome: Insulin in Blood
Description: A fasting blood sample was taken; insulin was quantified utilizing a commercial kit, that is based on the radioimmunoanalysis method (RIA).
Time Frame: At baseline and at months 1, 2, 3, 4, 5 and 6 of supplementation.
Measure: Median (Full Range); unit: µU/mL
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
µU/mL
  Basal | 10.2 [3.1 to 28.4] | 20.9 [3.0 to 49.2]
  Month 1 after supplement | 11.2 [5.5 to 38.5] | 17.8 [4.0 to 55.0]
  Month 2 after supplement | 12.2 [3.6 to 30.8] | 18.5 [2.4 to 50.0]
  Month 3 after supplement | 11.4 [3.2 to 34.1] | 18.0 [3.8 to 53.3]
  Month 4 after supplement | 9.2 [2.0 to 24.2] | 21.0 [3.9 to 60.0]
  Month 5 after supplement | 8.9 [2.3 to 25.9] | 17.7 [4.2 to 69.6]
  Month 6 after supplement | 10.6 [1.5 to 28.9] | 18.8 [1.9 to 61.6]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney) — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

6. Secondary Outcome: Inflammation Biomarkers (TNF-A)
Description: Plasma cytokine TNF-A was determined by enzyme-linked immunosorbent assay (ELISA) with a multiplex kit in picograms/mL.
Time Frame: Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Mean (Standard Deviation); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | 8.77 (50.01) | -1.45 (37.47)
  Month 2 after supplement | -22.04 (28.04) | -21.01 (37.69)
  Month 3 after supplement | -43.79 (32.69) | -37.76 (29.69)
  Month 6 after supplement | -65.78 (26.62) | -60.56 (18.77)
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority or Other; p > 0.05, Kruskal-Wallis — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

7. Secondary Outcome: Inflammation Biomarkers (IL-1)
Description: Plasma cytokine IL-1 was determined by enzyme-linked immunosorbent assay (ELISA) with a multiplex kit in picograms/mL.
Time Frame: Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Mean (Standard Deviation); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | 2.05 (53.77) | 21.74 (60.76)
  Month 2 after supplement | -6.00 (60.69) | -2.49 (76.14)
  Month 3 after supplement | -43.84 (34.96) | -9.89 (63.68)
  Month 6 after supplement | -57.04 (31.56) | -10.97 (70.95)
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p < 0.05, Kruskal-Wallis — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

8. Secondary Outcome: Inflammation Biomarkers (IL-6)
Description: Plasma cytokine IL-6 was determined by enzyme-linked immunosorbent assay (ELISA) with a multiplex kit in picograms/mL.
Time Frame: Time Frame: At baseline and at months 1, 2, 3, and 6 of supplementation.
Measure: Mean (Standard Deviation); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | 0.60 (43.80) | 0.08 (63.76)
  Month 2 after supplement | -10.57 (44.95) | -3.6 (41.66)
  Month 3 after supplement | -29.33 (35.17) | -16.61 (46.39)
  Month 6 after supplement | -52.33 (20.89) | -24.83 (48.15)
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

9. Secondary Outcome: Inflammation Biomarkers (IL-10)
Description: Plasma cytokine IL-10 was determined by enzyme-linked immunosorbent assay (ELISA) with a multiplex kit in picograms/mL.
Time Frame: Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Mean (Standard Deviation); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | 27.66 (115.80) | -8.89 (68.42)
  Month 2 after supplement | 4.83 (114.65) | -21.16 (50.03)
  Month 3 after supplement | 46.49 (171.49) | -39.91 (32.72)
  Month 6 after supplement | 108.85 (173.87) | -41.21 (52.60)
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p < 0.05, Kruskal-Wallis — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

10. Secondary Outcome: Inflammation Biomarker (IL-6 Expression)
Description: The messenger ribonucleic acid (mRNA) expression of cytokines IL-6 from circulating leucocytes was determined by quantifying the real-time polymerase chain reaction (PCR).
Time Frame: Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Mean (Standard Deviation); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Basal | 2.27 (2.7) | 2.45 (2.45)
  Month 1 after supplement | 1.26 (1.95) | 5.33 (4.47)
  Month 2 after supplement | 1.7 (0.88) | 7.82 (4.44)
  Month 3 after supplement | 0.6 (0.26) | 3.5 (2.72)
  Month 6 after supplement | 0.77 (0.39) | 9.5 (1.17)
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p < 0.05, t-test, 1 sided — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

11. Secondary Outcome: Inflammation Biomarker (TNF-A Expression)
Description: The messenger ribonucleic acid (mRNA) expression of cytokines TNF-A from circulating leucocytes was determined by quantifying the real-time polymerase chain reaction (PCR)
Time Frame: Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Mean (Standard Deviation); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Basal | 1.82 (2.6) | 1.15 (0.63)
  Month 1 after supplement | 2.07 (2.6) | 1.05 (0.94)
  Month 2 after supplement | 1.3 (2.07) | 2.12 (0.93)
  Month 3 after supplement | 1.05 (2.0) | 2.27 (3.11)
  Month 6 after supplement | 1.25 (1.43) | 0.52 (0.41)
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p < 0.05, t-test, 1 sided — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

12. Secondary Outcome: Inflammation Biomarker (IL-1 Expression)
Description: The messenger ribonucleic acid (mRNA) expression of cytokines IL-1 was determined by quantifying the real-time polymerase chain reaction (PCR).
Time Frame: Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Mean (Standard Deviation); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Basal | 1.22 (0.96) | 1.7 (1.78)
  Month 1 after supplement | 0.93 (1.24) | 1.08 (1.02)
  Month 2 after supplement | 0.69 (0.51) | 0.86 (0.41)
  Month 3 after supplement | 0.29 (0.16) | 0.66 (0.46)
  Month 6 after supplement | 0.47 (0.4) | 1.93 (0.87)
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p = 0.05, t-test, 1 sided — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

13. Secondary Outcome: Markers of Muscle Degeneration (Creatinine Kinase)
Description: The concentration in serum of CK was determined by chemiluminescent immunometric assay in U/L.
Time Frame: Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Mean (Standard Deviation); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | 23.30 (38.56) | 8.82 (52.59)
  Month 2 after supplement | 30.10 (58.23) | -9.95 (55.82)
  Month 3 after supplement | 8.45 (38.24) | 0.75 (44.76)
  Month 6 after supplement | 4.46 (42.67) | -1.52 (33.98)
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p > 0.05, Kruskal-Wallis — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

14. Secondary Outcome: Markers of Muscle Degeneration (MMP9)
Description: Plasma matrix metalloproteinase 9 (MMP9) was determined by enzyme-linked immunosorbent assay (ELISA) with a multiplex kit in ng/mL.
Time Frame: Time Frame: At baseline and at months 1, 2, 3 of supplementation.
Measure: Median (Full Range); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | -31.5 [-84.0 to 58.5] | -13.0 [-74.4 to 168.4]
  Month 2 after supplement | -3.5 [-58.8 to 315.6] | 47.7 [-73.0 to 274.2]
  Month 3 after supplement | -21.2 [-61.9 to 92.0] | 53.5 [-59.1 to 526.6]
  Month 6 after supplement | -23.6 [-58.0 to 37.3] | 39.9 [-40.1 to 443.0]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p > 0.05, Kruskal-Wallis — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

15. Secondary Outcome: Markers of Muscle Degeneration (sFas)
Description: The concentration in plasma of soluble Fas (sFas) was determined by enzyme-linked immunosorbent assay (ELISA) with a multiplex kit in picograms/mL.
Time Frame: Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Median (Full Range); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | 11.1 [-87.4 to 33.0] | 15.8 [-49.8 to 89.5]
  Month 2 after supplement | 14.2 [-89.0 to 53.5] | 15.8 [-29.7 to 67.2]
  Month 3 after supplement | 7.2 [-88.8 to 47.1] | 14.5 [-53.5 to 89.7]
  Month 6 after supplement | 18.3 [-89.5 to 157.7] | 20.7 [-34.7 to 51.2]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p > 0.05, Kruskal-Wallis — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

16. Secondary Outcome: Markers of Muscle Degeneration (Receptor of Fas)
Description: The concentration in plasma of the receptor o Fas (rFas) was determined by enzyme-linked immunosorbent assay (ELISA) with a multiplex kit in picograms/mL.
Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Median (Full Range); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | 16.5 [-45.3 to 95.7] | -2.0 [-62.5 to 5.0]
  Month 2 after supplement | 2.4 [-54.3 to 47.7] | -10.1 [-56.5 to 15.4]
  Month 3 after supplement | -15.7 [-44.2 to 28.8] | -16.3 [-58.5 to 49.7]
  Month 6 after supplement | -16.5 [-54.4 to 14.9] | -30.0 [-61.2 to 30.9]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority or Other; p > 0.05, Kruskal-Wallis — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

17. Secondary Outcome: Markers of Muscle Regeneration (VEGF)
Description: Vascular endothelial growth factor (VEGF) was quantified using enzyme linked immunosorbent assay (ELISA).
Time Frame: Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Median (Full Range); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | -25.9 [-89.6 to 75.3] | -5.7 [-75.3 to 182.1]
  Month 2 after supplement | 2.4 [-47.0 to 123.3] | -9.5 [-46.3 to 169.0]
  Month 3 after supplement | -15.7 [-44.2 to 28.8] | -16.3 [-58.5 to 49.7]
  Month 6 after supplement | -15.9 [-40.0 to 26.9] | 14.3 [-39.0 to 42.6]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p > 0.05, Kruskal-Wallis — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

18. Secondary Outcome: Markers of Muscle Regeneration (FGF)
Description: Plasma marker of regeneration fibroblast growth factor basic (FGF) was determined by enzyme-linked immunosorbent assay (ELISA) with a multiplex kit in picograms/mL.
Time Frame: Time Frame: At baseline and at months 1, 2, 3 and 6 of supplementation.
Measure: Median (Full Range); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | -13.6 [-76.2 to 133.6] | -37.3 [-79.7 to 50.2]
  Month 2 after supplement | 2.4 [-47.0 to 123.3] | -9.5 [-46.3 to 169.0]
  Month 3 after supplement | -0.92 [-69.8 to 186.2] | -57.1 [-89.2 to 81.9]
  Month 6 after supplement | -28.0 [-87.0 to 18.0] | -70.9 [-80.0 to 20.8]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p = 0.05, Kruskal-Wallis — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

19. Secondary Outcome: Incorporation of DHA in the Erythrocytes
Description: The percentage of DHA in the membrane of erythrocytes was determinated by gas chromatography.
Time Frame: Time Frame: At baseline and at months 1, 2, 3, 4, 5 and 6 of supplementation.
Measure: Median (Full Range); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | 57.8 [-34.4 to 721.9] | 0.9 [-79.0 to 77.2]
  Month 2 after supplement | 31.1 [-63.2 to 364.1] | -2.1 [-78.9 to 98.5]
  Month 3 after supplement | 153.4 [-43.7 to 1385.8] | -17.4 [-89.9 to 96.0]
  Month 4 after supplement | 247.6 [-49.5 to 1100.6] | 5.6 [-59.4 to 76.6]
  Month 5 after supplement | 116.6 [-35.2 to 1163.8] | -0.6 [-77.7 to 125.2]
  Month 6 after supplement | 289.4 [-82.7 to 2117.6] | -1.5 [-73.8 to 79.9]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

20. Secondary Outcome: Incorporation of EPA in the Erythrocytes
Description: The percentage of EPA in the membrane of erythrocytes was determinated by gas chromatography.
Time Frame: Time Frame: At baseline, at 1, 2, 3, 4, 5, and 6
Measure: Median (Full Range); unit: percentage of change respect at basal
Arm/Group | EPA and DHA | Sunflower Oil
Number analyzed (Participants) | 17 | 19
percentage of change respect at basal
  Month 1 after supplement | 233.0 [4.0 to 604.7] | -11.8 [-87.63 to 18.8]
  Month 2 after supplement | 300.4 [-10.7 to 656.3] | -11.5 [-87.6 to 274.0]
  Month 3 after supplement | 552.6 [168.6 to 1185.1] | -19.5 [-91.0 to 96.9]
  Month 4 after supplement | 552.7 [-86.7 to 999.3] | -20.9 [-80.2 to 14.4]
  Month 5 after supplement | 480.6 [23.4 to 2356.3] | -5.4 [-81.0 to 92.6]
  Month 6 after supplement | 446.4 [-51.8 to 1174.4] | -53.1 [-77.2 to 20.2]
Statistical Analysis 1: Comparison: EPA and DHA vs Sunflower Oil; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — Between-groups analysis (omega 3 vs placebo) at 3 and 6 months

ADVERSE EVENTS:
Time Frame: One patient presented vomiting and diarrhea, the patient had three evacuations during the night in a period of 3 hours and vomiting occurred for a period of 10 minutes. These complications occurred only once in the first month of supplementation.
Groups:
- EPA and DHA: Supplementation of 2.9 g / d of EPA and DHA will be provided in 10 capsules per day (4 in the morning, 3 in the afternoon and 3 at night) during a period of 6 months. The capsules sizes are specially for children to improved the feeding process and its presentation is in gelatin capsules. The supplement is purified fish oil with pharmaceutical grade.
  EPA and DHA: Each capsule contains 245mg of DHA, 45mg of EPA, other omega 3 50mg, oleic acid 60mg and Vitamin E 7.5 I. U.
- Sunflower Oil: Supplementation of placebo with sunflower fatty at doses of 10 capsules per day (4 in the morning, 3 in the afternoon and 3 at night) during a period of 6 months. The capsules sizes are specially for children to improved the feeding process. This placebo is sunflower oil and so will not expected to produce anti-inflammatory or insulin sensitivity effects.
  Placebo Comparator: Sunflower oil; the placebo capsules will also contain sunflower oil. Each gram contains: myristic (C14: 0 0) 1 mg, palmitic (C16: 0) 62mg, stearic (C18: 0) 43mg, palmitoleic (C16: 1) 1mg, oleic (C18: 1) 202mg, linolenic (C18: 3) 1mg and linoleic (C18: 2) 632mg.
Arm/Group | EPA and DHA | Sunflower Oil
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 1/18 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPA and DHA (N=18) | Sunflower Oil (N=22)
Vomiting and diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — One patient presented vomiting and diarrhea, the patient had three evacuations and one time of vomiting.

LIMITATIONS AND CAVEATS:
Limitations:

The sample size was not completed mainly because patients were not eligible for inclusion.

It was not possible to standardize the technical procedures for DNA fragmentation evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes